CLINICAL TRIAL: NCT04224753
Title: INVSENSOR00027 Fall Detection Clinical Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19817A
Record Dates: First submitted 2019-12-19; First posted 2020-01-13 (Actual); Results first posted 2020-06-01 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INVSENSOR00027 Test group (Experimental): The subjects will be enrolled into the test group and will receive the INVSENSOR00027 investigational sensor.
  Interventions: Device: INVSENSOR00027

INTERVENTIONS:
Device: INVSENSOR00027 — Investigational, noninvasive sensor that will be placed on the subject's chest. INVSENSOR00027 detects falls for each subject.

SUMMARY:
This study assesses INVSENSOR00027's clinical performance for fall detection.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old
* Physical status of ASA I or II
* Subjects must be able to read and communicate in English
* Has signed all necessary related documents, e.g. written informed consent, volunteer payment form, confidentiality agreement
* Has completed Health Assessment Questionnaire and passed health assessment screening

Exclusion Criteria:

* Subject has any medical condition which in the judgment of the investigator, renders them inappropriate for participation in this study
* Inability to tolerate physical activities including jumping and fall simulation
* Nursing female volunteers
* Excluded at the Principal Investigator's discretion
* Refusal to take the pregnancy test (for female subjects)
* Positive pregnancy test for female subjects of child bearing potential. This is done for the safety of this population.
* Refusal to shave hair (chest) off areas where sensors will be applied (male subjects)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Alghazi, Principal Investigator — Masimo Corporation
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00027 Test Group
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00027 Test Group
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 8
  Asian or Pacific Islander | 10
  Caucasian | 18
  Hispanic | 13
  Middle Eastern | 2
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of INVSENSOR00027's Fall Detection.
Description: For each subject's fall simulation, INVSENSOR00027 output will be computed. In order to calculate sensitivity of the device, true positives and false negatives need to be accounted for. For each event of fall, the sensor's output is observed. Fall that is correctly identified is marked as true positive (TP), whereas a missed detection is marked as false negative (FN). Combining the two, test sensitivity is computed by multiplying TP by 100 and dividing that over the sum of TP and FN.
Time Frame: 1-5 hours
Population: 1 subject excluded as study procedures were not followed per protocol.
Measure: Number; unit: percentage of falls detected
Arm/Group | INVSENSOR00027 Test Group
Number analyzed (Participants) | 50
percentage of falls detected | 93.9

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study (9 days).
Arm/Group | INVSENSOR00027 Test Group
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT04224753/Prot_SAP_000.pdf